CLINICAL TRIAL: NCT05418348
Title: A Phase 1, Randomized, Two-Period Crossover Study to Evaluate the Relative Bioavailability of Intravenous GTX-104 Compared to Oral Nimodipine Capsules at Steady State in Healthy Male and Female Subjects
Brief Title: Relative Bioavailability of Intravenous GTX-104 Compared to Oral Nimodipine Capsules in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grace Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GTX-104-002
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Nimodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (GTX-104 IV, Test): (Experimental): Nimodipine was administered by infusion over 72 hours.
  Interventions: Drug: GTX-104
- Treatment B (NIMOTOP, RLD): (Experimental): Nimodipine capsules (RS) administered orally with 240 mL of water at a dose level of 60 mg (two 30 mg capsules) q4h for 72 hours.
  Interventions: Drug: Nimodipine Capsules

INTERVENTIONS:
Drug: GTX-104 — new formulation of nimodipine injection for IV infusion
  Arms: Treatment A (GTX-104 IV, Test):
Drug: Nimodipine Capsules — Nimodipine capsules (reference formulation)
  Arms: Treatment B (NIMOTOP, RLD):

SUMMARY:
This is a Phase 1, single center, randomized, two-period crossover study in healthy male and female subjects designed to evaluate the relative bioavailability (BA) and safety at steady state of two formulations of nimodipine: GTX 104 (nimodipine for intravenous [IV] infusion; test formulation) and nimodipine oral capsules, RS (reference formulation).

ELIGIBILITY:
Inclusion Criteria:

* Subject had a body mass index between 18 and 32 kg/m2, inclusive.
* Subject was in good general physical health as determined by absence of clinically significant (CS) medical or psychiatric history, physical examination findings, vital signs, clinical laboratory evaluations, and 12-lead ECG measurements.

Exclusion Criteria:

* History or presence of clinically significant medical illness, including, but not limited to, cardiovascular, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic, psychiatric, renal, hepatic, chronic respiratory, or gastrointestinal disease, that could have interfered with the interpretation of the study.
* Had current or recent (within 6 months) history of gastrointestinal disease or any surgical or medical condition (eg, Crohn's or liver disease) that could potentially alter the absorption, metabolism, or excretion of the study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Cmax Day 1 | Day 1 for the first dose (8:00 AM dose)
  Maximum concentration
AUC (AUCDay 3, 0-24hr) | Day 3 from 8:00 AM to 8:00 AM from 0 to 24 hr
  Area under the concentration-time curve

SECONDARY OUTCOMES:
Cmax Day 3 across all 6 doses | Day 3
  Maximum concentration across all doses
Absolute bioavailability (F) Day 3 | Day 3
  the ratio of geometric LSmeans with corresponding 90% confidence interval calculated from the exponential of the difference between the Treatment-1 and Treatment-2 for the ln-transformed parameters Cmax Day3
Total body clearance of the drug from plasma after IV infusion (CL) Day 3 | Day 3 from 8:00 AM to 8:00 AM from 0 to 24 h
  (Dosedaily/AUCDay3,0-24)
Apparent total body clearance of the drug from plasma after oral administration (CL/F) Day 3 | Day 3 from 8:00 AM to 8:00 AM from 0 to 24 h
  Dosedaily/AUCDay 3 0-24

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Clinical Research Unit
Locations (1):
- Clinical Research Unit, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No